CLINICAL TRIAL: NCT05773079
Title: Toripalimab Maintenance After First-line Comprehensive Therapy for Locally Advanced Head and Neck Squamous Cell Carcinoma: a Single-arm, Phase II Study
Brief Title: Toripalimab Maintenance for Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2022-371
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma
Keywords: Squamous Cell Carcinoma of Head and Neck; Toripalimab; PFS; Immunotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab (Experimental): Toripalimab 240mg, VD, Q3W (treatment time: maintain for 1 year or until disease progression or intolerance requires drug withdrawal)
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Within 4 to 12 weeks after the first line of treatment, the maintenance treatment of Toripalimab was started, and 240 mg of Toripalimab was injected intravenously every 3 weeks (the maintenance treatment time was not more than 1 year, until there was an intolerable toxic reaction, or disease progression, or withdrawal of consent, or the investigator judged that it was necessary to withdraw from the treatment, or the subject had received treprizumab treatment for a cumulative period of 1 year or other reasons specified in the protocol). During the treatment period, tumor imaging evaluation shall be conducted every 3 months to see the research process description for details, and the evaluation shall be conducted according to the evaluation criteria of recist. If the evaluation is progress, the treatment shall be stopped.

SUMMARY:
The guidelines for locally advanced head and neck squamous cell carcinoma currently recommend surgery / radiotherapy / chemotherapy / targeted therapy. However, the median PFS of patients with high risk factors after comprehensive treatment was about 17 months, and the 2-year PFS rate was about 40 %. The KEYNOTE-048 study showed that PD-1 monoclonal antibody alone or in combination with chemotherapy significantly improved survival and was safe for recurrent / metastatic head and neck squamous cell carcinoma. Therefore, PD-1 monoclonal antibody has become the first-line treatment of metastatic head and neck squamous cell carcinoma. For locally advanced head and neck squamous cell carcinoma, the existing studies on immunotherapy for neoadjuvant or concurrent chemoradiotherapy have not been clearly concluded. We previously used PD-1 monoclonal antibody for the maintenance treatment of patients after the first-line treatment of locally advanced head and neck squamous cell carcinoma, without residual tumor, which showed a trend of prolonged survival. Therefore, this study intends to explore whether the maintenance treatment of PD-1 monoclonal antibody terripril can further improve the survival of patients with locally advanced head and neck squamous cell carcinoma with high risk factors and no residual tumor after first-line comprehensive treatment, and the safety is good.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced squamous cell carcinoma of the head and neck (AJCC8thIII-IV) confirmed by pathology in the initial treatment;
* No residual lesions after first-line surgery/radiotherapy/chemotherapy/targeted comprehensive treatment;
* Associated high risk factors: T3-4, regional lymph node positive, vascular invasion, neural invasion, lymph node capsular invasion, incisional margin positive;
* The patients' age is between 18 and 70 years old;
* The ECOG physical fitness status score is 0 or 1;
* Estimated survival period ≥ 3 months;
* The main organ functions meet the following standards: (1) Blood routine (without blood transfusion within 14 days): HGB ≥ 110g /L, WBC ≥ 3.0 × 10^9\/L， NEUT≥1.5 × 10^9\/L，PLT ≥75 × 10^9\/L； (2) Biochemical: BIL ≤ 1.5 times the upper limit of normal value (ULN), ALT and AST ≤ 2.0 × ULN, serum Cr ≤ 1.5 × ULN or endogenous creatinine clearance ≥ 50ml /min; (3) Occult blood in stool (-); (4) Normal urine routine, or urine protein<(++), or 24-hour urine protein<1.0g; (5) Left ventricular ejection fraction (LVEF) ≥ 50%. (6) The blood coagulation function is normal, and there is no active bleeding or thrombosis disease. A. International standardized ratio INR ≤ 1.5 × ULN； B. Partial thromboplastin time APTT ≤ 1.5 × ULN； C. Prothrombin time PT ≤ 1.5ULN. (7) Thyroid stimulating hormone (TSH) ≤ 1.5ULN; If the T3 and T4 levels are abnormal, they should be investigated. If the T3 and T4 levels are normal, they can be selected;
* Women of childbearing age should agree to use contraceptives (such as intrauterine devices, birth control pills, or condoms) during and within 3 months after the end of medication; "Within 7 days prior to study enrollment, the serum or urine pregnancy test was negative and must be a non lactating patient. The male should agree to use contraception during the study period and within 3 months after the end of the study period;
* Patients with hepatitis B virus (HBV) infection, inactive/asymptomatic HBV carriers, or patients with chronic or active HBV who received antiviral therapy for>1 week at the time of screening are allowed to be enrolled and continue treatment for more than 6 months after the study drug treatment. Patients with positive hepatitis C antibodies who have started anti hepatitis C virus treatment at the time of screening will be allowed to participate in the group;
* Subjects voluntarily joined the study, signed an informed consent form, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

* Distant metastasis of the tumor was detected upon enrollment;
* Have a history of allergy to PD-1 monoclonal antibody or drug components;
* There has been a history of other malignant tumors within the past 5 years or at the same time, except for cured skin basal cell carcinoma, cervical carcinoma in situ, and thyroid papillary carcinoma;
* Uncontrolled clinical cardiac symptoms or diseases, such as: (1) heart failure above NYHA class II; (2) unstable angina; (3) myocardial infarction within 1 year; (4) patients with clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention;
* Have received any of the following treatments: a. Have previously received treatment with immunosuppressive drugs; B. Have received any investigational drug within 4 weeks before the first use of the investigational drug; C. Joining another clinical study at the same time, unless it is an observational (non intervention) clinical study or an intervention clinical study follow-up; D. Subjects who require systemic treatment with corticosteroids (greater than 10 mg prednisone equivalent dose per day) or other immunosuppressants within 2 weeks prior to the first use of the study drug, excluding the use of corticosteroids for local inflammation and the prevention of allergies, nausea, and vomiting. In the absence of active autoimmune diseases, it is allowed to inhale or locally use steroids and adrenal cortical hormone replacement with a dose greater than 10 mg/day of prednisone; E. Have received an anti-tumor vaccine or a live vaccine within 4 weeks before the first administration of the study drug; F. Major surgery or severe trauma requiring removal of the disease within 4 weeks before the first use of the study drug;
* Serious infections (CTCAE greater than Level 2) occurred within 4 weeks before the first use of the study drug, such as severe pneumonia, intracranial infection, etc. that require hospitalization;
* Have a history of active autoimmune diseases and autoimmune diseases, but does not include autoimmune mediated hypothyroidism treated with stable doses of thyroid replacement hormone; Type I diabetes with a stable dose of insulin; Patients with vitiligo or recovered childhood asthma/allergies who do not require any intervention in adulthood;
* Have a history of immunodeficiency, including HIV testing positive, or have other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation and bone marrow transplantation;
* Have a history of interstitial lung disease and non infectious pneumonia;
* Patients who have a history of active pulmonary tuberculosis infection through medical history or CT examination, or who have a history of active pulmonary tuberculosis infection within 1 year before enrollment, or who have a history of active pulmonary tuberculosis infection before 1 year but have not received formal treatment;
* Subjects with active hepatitis (HBV DNA ≥ 2000 IU /ml or 10000 copies /ml) who have not been treated, and hepatitis C (hepatitis C antibody positive, and HCV-RNA above the detection limit of the analytical method) who have not been treated;
* Known history of abuse, alcoholism, and drug abuse of psychotropic substances;
* KPS score<60, intolerance to anti-tumor therapy;
* Pregnant or lactating women;
* Engaging or expected to participate in other clinical studies;
* Researchers believe that it is not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival | 2 years
  The time from the day of first-line systemic treatment to disease progression or death.

SECONDARY OUTCOMES:
2-year Overall Survival | 2 years
  The time from the day of first-line treatment to the death of any cause.

OTHER OUTCOMES:
≥Grade 3 Treatment-Related Adverse Events | 2 years
  Any adverse signs ( including abnormal laboratory results ), symptoms or diseases that are time-related to the use of the study drug, regardless of whether there is a causal relationship with the study drug